CLINICAL TRIAL: NCT02501421
Title: Reactogenicity, Safety and Immunogenicity of a TB/FLU-04L Tuberculosis Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Research Institute for Biological Safety Problems (Other Government)
Collaborators: Ministry of Health, Kazakhstan (Other Government); Research Institute of Influenza, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VPT-I-01/2013
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2015-07

CONDITIONS: Tuberculosis
Keywords: vaccine; influenza vector; tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Tuberculosis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TB/FLU-04L (Active Comparator): Live recombinant influenza vectored tuberculosis vaccine
  Interventions: Biological: tuberculosis vaccine
- Placebo (Placebo Comparator): Buffer
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: tuberculosis vaccine — Live recombinant influenza vectored tuberculosis vaccine
  Other Names: TB/FLU-04L
  Arms: TB/FLU-04L
Biological: Placebo — Buffer
  Arms: Placebo

SUMMARY:
The study is a single centre, phase I, double-blind, randomized, placebo-controlled trial that explored the safety and immunogenicity of 2 doses (Day 1 and Day 21) TB/FLU-04L tuberculosis vaccine versus matched placebo in BCG-vaccinated healthy adult subjects aged 18-50 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy BCG-vaccinated male or female adult 18 through 50 years of age at the enrollment visit.
* Literate and willing to provide written informed consent.
* A signed informed consent.
* Capable and willing to complete diary cards and willing to return for all follow-up visits.
* For females, willing to take reliable birth control measures throughout the entire period of participation in the study.

Exclusion Criteria:

* Clinical, radiological (chest X-ray) or laboratory evidence of active or past TB disease.
* Current or past administration of anti-TB therapy.
* History of contact with TB patients.
* Positive QuantiFERON-TB Gold test.
* BCG vaccination in less than 6 months prior to study.
* Practice of nasal irrigation on a regular basis within the past six months or has engaged in nasal irrigation within two weeks prior to enrollment.
* Recent history of frequent nose bleeds (>5 within the past year).
* Clinically relevant abnormal paranasal anatomy.
* Recent history (within the past month) of rhino or sinus surgery, or surgery for any traumatic injury of the nose.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Hypersensitivity after previous administration of any vaccine.
* History of chronic alcohol abuse and/or illegal drug use.
* Any clinically significant abnormal laboratory finding.
* A positive pregnancy test for all women of childbearing potential.
* Administration of immunosuppressive drugs or other immune modifying drugs within 4 weeks prior to study enrollment.
* Acute or chronic clinically significant pulmonary disease, cardiovascular disease, gastrointestinal disease, liver disease, neurological illness, liver disease, blood disease, skin disorder, endocrine disorder, neurological illness and psychiatric disorder as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives.
* History of leukemia or any other blood or solid organ cancer.
* Seropositive for HIV, hepatitis B surface antigen and/or hepatitis C antibodies.
* Receipt of antivirals, antibiotics, immunoglobulins or other blood products within 4 weeks prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Participation in another clinical trial within the previous three months or planned enrollment in such a trial during the period of this study.
* Subjects who are, in the opinion of the investigator, at significantly increased risk of non-cooperation with requirements of the study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Immediate reactions | Two hours
  Immediate reactions occurring within two hours of administration of any dose
Solicited local and systemic reactions | Greater than 2 hours after administration of any dose of vaccine or placebo through 7 days following any dose
  Adverse events commonly associated with intranasal vaccination
Unsolicited events and abnormal laboratory findings | Greater than 2 hours after administration of any dose of vaccine or placebo through 7 days following any dose
  Adverse events not associated with intranasal vaccination and abnormal laboratory findings
Serious adverse events (SAEs), including abnormal laboratory findings | Three weeks of receipt of any dose
  All SAEs during three weeks after receipt of any dose